CLINICAL TRIAL: NCT01426295
Title: Pharmaco-economic Cost-effective Prospective Randomized Trial Evaluating the Open Interest Caphosol ® Mouthwashes in the Prevention and Treatment of Severe Oral Mucositis in Patients Receiving High-dose Chemotherapy in Hematology
Brief Title: Pharmaco-economic Study of a New Medical Device Performed From the Perspective of the Hospital
Acronym: Caphosol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: BRD/10/06-C
Record Dates: First submitted 2011-08-26; First posted 2011-08-31 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Hematologic Disease
Keywords: hematologic disease candidates for autologous or allogeneic bone marrow
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Caphosol (Experimental)
  Interventions: Device: Caphosol
- Référence (Active Comparator): •Bicarbonate de sodium à 1.4% Biosedra Versylène® or PAROEX® :
  Interventions: Drug: Bicarbonate de sodium

INTERVENTIONS:
Device: Caphosol — The Caphosol ™ is a recently launched medical in France (2009). (source: laboratory EUSA Pharma ®)
  The product is an aqueous solution for mouthwash that comes in the form of a hyper-saturated mixture of calcium phosphate at neutral pH to reconstitute immediately before use.
  Each patient randomized to the treatment arms in the study will receive daily at least 4 (maximum 10) mouthwash Caphosol ™.
  The treatments are to begin preventive J1 to chemotherapy and continued until out of aplasia (ANC> 500/mm3), and / or mucositis grade 0.
  Arms: Caphosol
Drug: Bicarbonate de sodium — Treatment of the early start on the day of conditioning and stop when the ANC> 500/mm3 and / or mucositis grade zero, provisional date of bone exceeded.
  Versylène: Method of administration: gargle made with a minute from 15 to 30 mL, 2-5 times a day, alternating with PAROEX ®.
  Arms: Référence

SUMMARY:
The purpose of the study is to determine whether the use of mouthwashes Caphosol ™ in addition to standard oral care (strategy A) is cost-effective in the prevention and treatment of severe mucositis in adult patients with auto or allograft packaging without ICT versus mouthwashes standard bicarbonates with an antiseptic (strategy B).

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years

Patient receiving:

* Conditioning of autologous bone marrow transplantation by high dose melphalan (HD) as part of the management of myeloma or BEAM in lymphoma.
* A conditioning allogeneic bone marrow transplantation with reduced or intermediate busulfan IV
* Patients belong to a schema of social security, having signed the written informed consent.

Exclusion Criteria:

* patients:
* To receive or have received KGF
* With previous history of RT with the exception of patients who received spinal analgesic therapy in the treatment of myeloma
* Unable or unwilling to complete the self assessment questionnaire
* With previous history of allergy to any component of the products under consideration
* Minor
* Adults under guardianship
* Pregnant women
* Patients who have not signed the consent form
* Creation of mouthwash out of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2011-04; Primary Completion 2013-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
assess the cost-effectiveness ratio is the number of days with severe mucositis won. | up to 28 days

SECONDARY OUTCOMES:
The number of days without medication morphine won | up to 28 days
Aggregate saving medicines prescribed Supportive | up to 28 days
The incidence of mucositis | up to 28 days
The intensity of pain assessed with a visual analogue scale | up to 28 days
The cumulative dose of morphine administered and the number of days of treatment, | 28 days
The duration of febrile neutropenia | up to 28 days
- The incidence and duration of treatment of anti-infective and antifungal | 28 jours
The incidence of total parenteral nutrition | up to 28 days
- The duration of Release aplasia (ANC> 500/mm3), | up to 28 days
The duration of the hospitalization | participants will be followed for the duration of hospital stay, an expected average of 28 days
The severity of mucositis | up to 28 days
The duration of pain assessed with a visual analogue scale, | up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gastinne, M D, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes Universty Hospital, Nantes, France